CLINICAL TRIAL: NCT06491901
Title: Prospective, Non-Blinded, Randomized Controlled Trial on Early Administration of Pulmonary Surfactant Guided by Lung Ultrasound Scores in Very Preterm Infants.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2023337; M22018 (Other Grant/Funding Number: Beijing Natural Science Foundation)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Early Administration of Pulmonary Surfactant Guided by Lung Ultrasound Scores in Very Preterm Infants

STUDY DESIGN:
Intervention Model Description: A prospective, non-blinded, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): Lung ultrasonography will be performed within 1 h of admission, followed by lung ultrasound scoring.
  Interventions: Other: PS was given according to lung ultrasound score
- Control group (Active Comparator): NRDS was diagnosed according to clinical criteria.
  Interventions: Other: PS was given according to clinical criteria

INTERVENTIONS:
Other: PS was given according to lung ultrasound score — If the lung ultrasound confirms RDS and LUS is more than 8, a full dose of PS will be promptly administered at 200 mg/kg (Poractant Alfa, Curosurf®). If the lung ultrasound does not indicate RDS or if LUS is 8 or less, clinical monitoring will continue. Should the clinical criteria for NRDS be met, a full dose of PS will be administered at 200 mg/kg (Poractant Alfa, Curosurf®). In terms of the administration method, less-invasive surfactant administration (LISA) will be employed for infants in a non-invasive ventilation state, while those in an invasive ventilation state will receive PS via endotracheal tube.
  Arms: Ultrasound group
Other: PS was given according to clinical criteria — In cases where clinical diagnosis confirms NRDS, PS will be administered at a dosage of 200 mg/kg (Poractant Alfa, Curosurf®). LISA will be employed for infants in a non-invasive ventilation state, while those in an invasive ventilation state will receive PS via endotracheal tube. If clinical manifestations do not meet the diagnosis of NRDS, PS will not be administered.
  Arms: Control group

SUMMARY:
Abstract Background: Bedside lung ultrasonography has been widely used in neonatal intensive care units (NICUs). Lung ultrasound scores (LUS) may predict the need for pulmonary surfactant (PS) application. PS replacement therapy is the key intervention for managing moderate to severe neonatal respiratory distress syndrome (NRDS), with early PS administration playing a positive role in improving patient outcomes. Lung ultrasonography aids in the prompt diagnosis of NRDS, while LUS offers a semi-quantitative assessment of lung health. However, the specific methodologies for utilizing LUS in clinical practice remain controversial. This study hypothesizes that, in very preterm infants (<32 weeks gestational age [GA]) exhibiting respiratory distress symptoms, determining PS application through early postnatal LUS combined with clinical indicators, as opposed to relying solely on clinical signs and chest X-rays, can lead to more timely PS administration, reduce mechanical ventilation duration, improve patient outcomes, and lower the occurrence of bronchopulmonary dysplasia (BPD).

Methods and design: This is a protocol for a prospective, non-blinded, randomized controlled trial that will be conducted in the NICU of a hospital in China. Eligible participants will include very preterm infants (< 32 weeks GA) exhibiting signs of respiratory distress. Infants will be randomly assigned in a 1:1 ratio to either the ultrasound or control group. In the ultrasonography group, the decision regarding PS administration will be based on a combination of lung ultrasonography and clinical manifestations, whereas in the control group, it will be determined solely by clinical signs and chest X-rays. The primary outcome measure will be the mechanical ventilation duration. Statistical analysis will employ independent sample t-tests with a significance level set at α = 0.05 and a power of 80%. The study requires 30 infants per group (in total 60 infants).

Hypothesis: This study aims to demonstrate that determining PS application based on a combination of LUS and clinical indicators is superior to traditional approaches.

This approach may enhance the accuracy of NRDS diagnosis and facilitate early prediction of PS requirements, thereby reducing the duration of mechanical ventilation. The findings of this research may contribute valuable insights into the use of LUS to guide PS administration.

DETAILED DESCRIPTION:
Ultrasound group: Lung ultrasonography will be performed within 1 h of admission, followed by lung ultrasound scoring. If the lung ultrasound confirms RDS and LUS is more than 8, a full dose of PS will be promptly administered at 200 mg/kg (Poractant Alfa, Curosurf®). If the lung ultrasound does not indicate RDS or if LUS is 8 or less, clinical monitoring will continue. Should the clinical criteria for NRDS be met, a full dose of PS will be administered at 200 mg/kg (Poractant Alfa, Curosurf®). Lung ultrasound and scoring will be repeated 4 to 10 h post the first PS dose administration. Repeated PS administration will occur if the criteria are met, with lung ultrasound scoring conducted prior to each administration.

Control group: In cases where clinical diagnosis confirms NRDS, PS will be administered at a dosage of 200 mg/kg (Poractant Alfa, Curosurf®). If clinical manifestations do not meet the diagnosis of NRDS, PS will not be administered.

All enrolled infants will undergo lung ultrasound scoring at 24 h, 3 days, 7 days, 14 days, 28 days, and 36 weeks CA (prior to discharge).

ELIGIBILITY:
Inclusion Criteria:

Infants who meet all of the following criteria will be included: (1) very preterm infants with a GA of less than 32 weeks; (2) presence of respiratory distress after birth, such as a respiratory rate of more than 60 breaths/min, grunting, nasal flaring, intercostal retractions, and/or cyanosis; (3) born in the authors' hospital.

Exclusion Criteria:

Infants who meet any of the following criteria will be excluded: (1) infants who have received PS treatment in the delivery room or external setting after birth; (2) infants with known or confirmed congenital abnormalities, especially cardiopulmonary deformities during diagnosis or treatment; (3) presence of severe complications at birth (severe asphyxia, hemorrhagic shock, pneumonia, pneumothorax, early-onset sepsis, and pleural effusion) or other diseases not caused by PS deficiency; (4) infants who die within 72 h after birth, are transferred to another hospital for surgery, or have incomplete data; and (5) those with families who do not consent to participate in this study.

Ages: 10 Minutes to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
the duration of mechanical ventilation | At 36 weeks PMA or at discharge, whichever came first
  The duration of mechanical ventilation (both invasive and non-invasive) during hospitalization in the ultrasound and control groups.

SECONDARY OUTCOMES:
the utilization rate of PS | Within the first week of life
  The utilization rate of PS in both groups
the proportion of infants receiving the first dose of PS early | Within the first week of life
  The proportion of infants receiving the first dose of PS early (within 3 h after birth) and the time from birth to the initial PS administration
the worst oxygenation index (OI) | Within the first week of life
  The worst oxygenation index (OI) at different time points following PS administration
Lung Ultrasound Scores (LUS) | At 36 weeks PMA or at discharge, whichever came first
  LUS at various intervals following PS administration (at 3 days, 7 days, 14 days, 28 days, and before discharge/at 36 weeks CA)
Preterm comorbidities | At 36 weeks PMA or at discharge, whichever came first
  The incidence rates of major complications in preterm infants such as BPD, intraventricular hemorrhage (IVH), retinopathy of prematurity (ROP), and necrotizing enterocolitis (NEC)

IPD SHARING:
Plan to Share IPD: Undecided